CLINICAL TRIAL: NCT05571748
Title: The Association Between Oxidative Stress and Carbohydrate Metabolism Disorders in G6PD Deficient Individuals
Brief Title: Oxidative Stress, Carbohydrate Metabolism Disorders and G6PD Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Principal Investigator, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G6PD_Diabetes
Record Dates: First submitted 2022-05-28; First posted 2022-10-07 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: G6PD Deficiency; Carbohydrate Metabolism Disorder; Oxidative Stress
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency | interventions — Thioctic Acid; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- G6PD deficiency (only) - Intervention (Experimental): Alpha-lipoic acid supplementation (600 mg/day) for 4 weeks in a counterbalanced manner to 10 G6PD deficient individuals.
  Interventions: Dietary Supplement: Alpha-lipoic acid
- G6PD deficiency (only) - Placebo (Placebo Comparator): Placebo administration for 4 weeks in a counterbalanced manner to 120 G6PD deficient individuals.
  Interventions: Other: Placebo
- G6PD deficiency and CHO metabolism disorder - Intervention (Experimental): Alpha-lipoic acid supplementation (600 mg/day) for 4 weeks in a counterbalanced manner to 10 individuals with G6PD deficiency and a CHO metabolism disorder.
  Interventions: Dietary Supplement: Alpha-lipoic acid
- G6PD deficiency and CHO metabolism disorder - Placebo (Placebo Comparator): Placebo for 4 weeks in a counterbalanced manner to 10 individuals with G6PD deficiency and a CHO metabolism disorder.
  Interventions: Other: Placebo
- CHO metabolism disorder (only) - Intervention (Experimental): Alpha-lipoic acid supplementation (600 mg/day) for 4 weeks in a counterbalanced manner to 10 individuals with a CHO metabolism disorder.
  Interventions: Dietary Supplement: Alpha-lipoic acid
- CHO metabolism disorder (only) - Placebo (Placebo Comparator): Placebo for 4 weeks in a counterbalanced manner to 10 individuals with a CHO metabolism disorder.
  Interventions: Other: Placebo
- Controls - Intervention (Experimental): Alpha-lipoic acid supplementation (600 mg/day) for 4 weeks in a counterbalanced manner to 10 individuals without G6PD deficiency and/or any CHO metabolism disorder.
  Interventions: Dietary Supplement: Alpha-lipoic acid
- Controls - Placebo (Placebo Comparator): Placebo for 4 weeks in a counterbalanced manner to 10 individuals without G6PD deficiency and/or any CHO metabolism disorder.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Alpha-lipoic acid — A trial of acute exercise before and after 4 weeks of alpha-lipoic acid supplementation.
  Other Names: Physical exercise
  Arms: CHO metabolism disorder (only) - Intervention; Controls - Intervention; G6PD deficiency (only) - Intervention; G6PD deficiency and CHO metabolism disorder - Intervention
Other: Placebo — A trial of acute exercise before and after 4 weeks of placebo supplementation.
  Other Names: Physical exercise
  Arms: CHO metabolism disorder (only) - Placebo; Controls - Placebo; G6PD deficiency (only) - Placebo; G6PD deficiency and CHO metabolism disorder - Placebo

SUMMARY:
The purpose of this study is to investigate the effects of alpha-lipoic acid supplementation on redox status, physiological and biochemical parameters in diabetic individuals with G6PD deficiency, after acute exercise.

DETAILED DESCRIPTION:
In a randomized double-blind, crossover design, a total of forty people will participate in the research voluntarily: (a) ten people with G6PD (Mediterranean type) enzyme deficiency), (b) ten people with G6PD (Mediterranean type) enzyme deficiency and a disorder of carbohydrate metabolism (diabetes, prediabetes), (c) ten people with a disorder of carbohydrate metabolism (diabetes mellitus and prediabetes) and, (d) ten people without any health problem (control group). They will be supplemented with either 600 mg of alpha-lipoic acid (experimental condition) or placebo (control condition) every day for 4 weeks, separated by a 4-week washout period. All participants will be randomly assigned to both conditions.

Before intervention, all participants will be informed about the study protocol, fill a medical history questionnaire and sign an informed consent form. Moreover, measurements of anthropometric characteristics and physiological parameters, as well as a VO2peak test will be performed.

Participants will perform a trial of exercise (70% VO2peak for 45min and 90% till exhaustion) before and after each condition (i.e. a total of 4 trials). Blood samples will be collected before, immediately after and 1 hour after each exercise trial. Moreover, measurements of anthropometric characteristics, physiological and psychological parameters will be performed before and after each condition.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with normal G6PD activity
* Individuals with G6PD deficiency
* Individuals with CHO metabolism disorders (diabetes, prediabetes)
* Individuals with G6PD deficiency and CHO metabolism disorders (diabetes, prediabetes)

Exclusion Criteria:

* Health problems that contraindicate participation to exercise
* Should not take any medication that affects the body's antioxidant mechanisms as well as dietary supplements containing antioxidants
* Women during lactation or gestation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Changes in total antioxidant capacity following 4 weeks of supplementation and placebo at rest and following a trial of acute exercise. | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Index of blood redox status. Spectrophotometric assay for the determination of total antioxidant capacity using DPPH method.
Changes in glutathione following 4 weeks of supplementation and placebo at rest and following a trial of acute exercise. | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Index of blood redox status. Spectrophotometric assay for the determination of total antioxidant capacity using DTNB method.
Changes in uric acid following 4 weeks of supplementation and placebo at rest and following a trial of acute exercise. | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Index of blood redox status. Spectrophotometric assay for the determination of total antioxidant capacity using a clinical chemistry analyzer with commercially available kits.
Changes in bilirubin following 4 weeks of supplementation and placebo at rest and following a trial of acute exercise. | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Index of blood redox status. Spectrophotometric assay for the determination of bilirubin using a clinical chemistry analyzer with commercially available kits.
Changes in lipid peroxidation following 4 weeks of supplementation and placebo at rest and following a trial of acute exercise. | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Index of blood redox status. Determination of lipid peroxidation using malondialdehyde production assessment.
Changes in protein carbonyls following 4 weeks of supplementation and placebo at rest and following a trial of acute exercise. | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Index of blood redox status. Spectrophotometric assay for the determination of total antioxidant capacity using DNPH method.
Changes in blood lipids following 4 weeks of supplementation and placebo at rest and following a trial of acute exercise. | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Blood lipids (total cholesterol, LDL-c, HDH-c, triglycerides). Spectrophotometric assays for the determination of blood lipids using a clinical chemistry analyzer with commercially available kits.
Changes in insulin resistance following 4 weeks of supplementation and placebo. | Before and following 4 weeks of supplementation and placebo.
  Measurement of blood glucose and insulin levels to assess HOMA-IR and evaluate insulin resistance. Spectrophotometric assay for the determination of blood glucose using a clinical chemistry analyzer with commercially available kits.Determination of blood insulin using commercially available Eliza kits.
Changes in glycated hemoglobin (HbA1c) following 4 weeks of supplementation and placebo. | Before and following 4 weeks of supplementation and placebo.
  Measurement of HbA1c using commercially available kits.

SECONDARY OUTCOMES:
Changes in body composition following 4 weeks of intervention and placebo. | Before and following 4 weeks of supplementation and placebo.
  Body fat mass (in kg) and percentage, lean mass (in kg) and percentage
Changes in body mass index following 4 weeks of intervention and placebo. | Before and following 4 weeks of supplementation and placebo.
  Body mass (in kg) and height (in cm)
Changes in resting heart rate following 4 weeks of intervention and placebo. | Before and following 4 weeks of supplementation and placebo.
  Resting heart rate (beats per minute) measurement after at least 5 minutes at rest
Changes in blood pressure following 4 weeks of intervention and placebo. | Before and following 4 weeks of supplementation and placebo.
  Measurement of (systolic and diastolic) blood pressure (in mm Hg) after at least 5 minutes at rest
Changes in waist-to-hip ratio following 4 weeks of intervention and placebo. | Before and following 4 weeks of supplementation and placebo.
  Measurement of waist and hip circumference to calculate waist-to-hip ratio
Changes in complete blood count following 4 weeks of intervention and placebo. | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Complete blood count
Changes in psychometric test following 4 weeks of intervention and placebo. | Before and following 4 weeks of supplementation and placebo.
  Hospital Anxiety Depression Scale-HADS (Greek version)
Trial of VO2peak estimation. | Before intervention.
  VO2peak (mL/kg body weight/min) estimation with a treadmill protocol.
Nicotinamide-adenine dinucleotide phosphate (NADPH) | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Spectrophotometric assay for the determination of NADPH in erythrocytes.
Glutathione Reductase (GR) | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Spectrophotometric assay for the determination of GR in erythrocytes.
Glutathione peroxidase (GPx) | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Spectrophotometric assay for the determination of GPx in erythrocytes.
Superoxide dismutases (SOD) | Before, immediately after and 1 hour after each trial of exercise, in both conditions (supplement and placebo)
  Spectrophotometric assay for the determination of SOD in erythrocytes.
Glucose Tolerance Test (GTT) | Before intervention (blood samples at 0, 30, 60, 90 and 120 minutes after intake of 75 g glucose).
  GTT for the investigation of changes in glucose control.
G6PD enzyme activity in erythrocytes | Before intervention. During GTT (blood samples at 0, 30, 60, 90 and 120 minutes after intake of 75 g glucose). Also before, immediately after and 1, 2, 24 hours after each trial of exercise, in both conditions (supplement and placebo).
  Quantification of G6PD activity in erythrocytes (units/gram of hemoglobin) of all participants using a commercially available kit.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z Jamurtas, PhD, Study Director — University of Thessaly

REFERENCES:
- [Background] Georgakouli K, Deli CK, Zalavras A, Fatouros IG, Kouretas D, Koutedakis Y, Jamurtas AZ. Alpha-lipoic acid supplementation up-regulates antioxidant capacity in adults with G6PD deficiency. Food Chem Toxicol. 2013 Nov;61:69-73. doi: 10.1016/j.fct.2013.01.055. Epub 2013 Feb 14. PMID 23416142